CLINICAL TRIAL: NCT03691649
Title: A Phase III, Randomized, Double-Masked, Active-Controlled, Parallel-Group, Multi-center Study Assessing the Efficacy and Safety of DE-117 Ophthalmic Solution Compared With Timolol Maleate Ophthalmic Solution 0.5% in Subjects With Glaucoma or Ocular Hypertension - Spectrum 3 Study
Brief Title: A Phase III Study Assessing the Efficacy and Safety of DE-117 Ophthalmic Solution Compared With Timolol Maleate Ophthalmic Solution 0.5% in Subjects With Glaucoma or Ocular Hypertension - Spectrum 3 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 011709IN
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Results first posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Glaucoma and Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DE-117 Ophthalmic Solution (Experimental): Topical DE-117 Ophthalmic Solution once daily and Vehicle once daily for 3 months for all subjects, followed by DE-117 Ophthalmic Solution once daily for additional 9 month for adult subjects only
  Interventions: Drug: DE-117 Ophthalmic Solution
- Timolol Maleate Ophthalmic Solution 0.5% (Active Comparator): Topical Timolol Maleate Ophthalmic Solution 0.5% twice daily for 3 months for all subjects, followed by DE-117 Ophthalmic Solution once daily for additional 9 month for adult subjects only
  Interventions: Drug: Timolol Maleate Ophthalmic Solution 0.5%

INTERVENTIONS:
Drug: DE-117 Ophthalmic Solution — Topical DE-117 Ophthalmic Solution once daily and Vehicle once daily for 3 months for all subjects, followed by DE-117 Ophthalmic Solution once daily for additional 9 month for adult subjects only
  Arms: DE-117 Ophthalmic Solution
Drug: Timolol Maleate Ophthalmic Solution 0.5% — Topical Timolol Maleate Ophthalmic Solution 0.5% twice daily for 3 months for all subjects, followed by DE-117 Ophthalmic Solution once daily for additional 9 month for adult subjects only
  Arms: Timolol Maleate Ophthalmic Solution 0.5%

SUMMARY:
This is a Phase III, randomized, double-masked, active-controlled, parallel-group, multi-center study. Subjects diagnosed with glaucoma or OHT who meet eligibility criteria at Visit 1 (Screening) will washout of their current topical IOP-lowering medication(s), if any. After completing the required washout period, subjects will return for Visit 2 (Baseline, Day 1). Subjects who meet all eligibility criteria at baseline will be randomized to receive double-masked treatment for 3 months. Adult subjects will receive open-label DE-117 Ophthalmic Solution for an additional 9 months.

Approximately 400 adult subjects and up to 30 pediatric subjects with glaucoma or OHT who meet all eligibility criteria will be randomized in a 1:1 ratio to receive either:

* DE-117 Ophthalmic Solution once daily and Vehicle once daily, or
* Timolol Maleate Ophthalmic Solution 0.5% twice daily. The study will evaluate the efficacy and safety of DE-117 Ophthalmic Solution compared with Timolol Maleate Ophthalmic Solution 0.5% in subjects with glaucoma or OHT through Month 3 and will provide additional safety data through Month 12 for subjects receiving DE-117.

ELIGIBILITY:
Inclusion Criteria:

• glaucoma or ocular hypertension

Exclusion Criteria:

* Females who are pregnant, nursing, or planning a pregnancy
* Any corneal abnormality or other condition interfering with or preventing reliable tonometric measurements

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-09-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (47):
- United States (47):
  - Arizona Glaucoma Specialists, Phoenix, Arizona
  - DocTrials Walman Eye Center, Sun City, Arizona
  - Havana Research Institute, Burbank, California
  - Macy Eye Center, Los Angeles, California
  - North Valley Eye Medical Group, Mission Hills, California
  - North Bay Eye Associates, Inc, Petaluma, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Samsum Clinic (DocTrials), Santa Barbara, California
  - MCB Clinical Research Centers LLC, Colorado Springs, Colorado
  - Hernando Eye Institute, Brooksville, Florida
  - Eye Associates of Fort Myers, Fort Myers, Florida
  - Bowden Eye & Associates, Jacksonville, Florida
  - Shettle Eye Research, Largo, Florida
  - Dixophthal PC Dba. Dixon Eye Care, Albany, Georgia
  - Coastal Research Associates, Alpharetta, Georgia
  - Clayton Eye Clinical Research, LLC, Morrow, Georgia
  - Indiana University, Bloomington, Indiana
  - Heart of America Eye Care, P.A., Shawnee Mission, Kansas
  - Clinical Eye Research of Boston, LLC, Winchester, Massachusetts
  - Tauber Eye Center, Kansas City, Missouri
  - Nevada Eye Care Professionals, Las Vegas, Nevada
  - Wellish Vision Institute, Las Vegas, Nevada
  - AdvanceMed Clinical Research-Las Vegas, Las Vegas, Nevada
  - Northern New Jersey Eye Institute, South Orange, New Jersey
  - NY Eye & ear Infirmary of Mt Sinai (NYEE), New York, New York
  - South Shore Eye Care, LLP, Wantagh, New York
  - Asheville Eye Associates, Asheville, North Carolina
  - Charlotte Eye Ear Nose & Throat Associates, PA, Charlotte, North Carolina
  - Cornerstone Eye Care, High Point, North Carolina
  - Apex Eye Clinical Research, LLC, Cincinnati, Ohio
  - Ophthalmic Surgeons & Consultants of Ohio, Inc., Columbus, Ohio
  - Office of Mark J. Weiss MD, Tulsa, Oklahoma
  - Scott & Christie and Associates PC, Cranberry Township, Pennsylvania
  - Glaucoma Consultants and Center for Eye Research PA, Mt. Pleasant, South Carolina
  - Black Hills Regional Eye Institute, LLP, Rapid City, South Dakota
  - University Eye Specialists, Maryville, Tennessee
  - Total Eye Care PA, Memphis, Tennessee
  - Keystone Research Ltd. Texan Eye PA, Austin, Texas
  - The Cataract and Glaucoma Center, El Paso, Texas
  - Ophthalmology Associates, Fort Worth, Texas
  - Shah Research LLC dba Discovery Clinical Trials, Mission, Texas
  - San Antonio Eye Center, San Antonio, Texas
  - R and R Eye Research LLC, San Antonio, Texas
  - Delay Winter Eye Consultants LLC, San Antonio, Texas
  - Stacy R. Smith M.D. P.C., Salt Lake City, Utah
  - Emerson Clinical Research Institute, Falls Church, Virginia
  - Specialty Eye Care Centre, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DE-117 Ophthalmic Solution: Topical DE-117 Ophthalmic Solution once daily and Vehicle once daily for 3 months for all subjects, followed by DE-117 Ophthalmic Solution once daily for additional 9 months for adult subjects only.
  DE-117 Ophthalmic Solution: Topical DE-117 Ophthalmic Solution once daily and Vehicle once daily for 3 months for all subjects, followed by DE-117 Ophthalmic Solution once daily for additional 9 months for adult subjects only.
- Timolol Maleate Ophthalmic Solution 0.5%: Topical Timolol Maleate Ophthalmic Solution 0.5% twice daily for 3 months for all subjects, followed by DE-117 Ophthalmic Solution once daily for additional 9 months for adult subjects only.
  Timolol Maleate Ophthalmic Solution 0.5%: Topical Timolol Maleate Ophthalmic Solution 0.5% twice daily for 3 months for all subjects, followed by DE-117 Ophthalmic Solution once daily for additional 9 months for adult subjects only.
Period: Double Masked Treatment Period (DMTP)
Arm/Group | DE-117 Ophthalmic Solution | Timolol Maleate Ophthalmic Solution 0.5%
Started | 212 (Includes 6 pediatric participants.) | 214 (Includes 7 pediatric participants.)
Full Analysis Set Participants | 212 | 213
Safety Analysis Set Participants | 211 (One participant that was randomized to DE-117 arm inadvertently received Timolol during Double Masked Treatment Period hence 211 participants were dosed with study drug and assessed for safety.) | 215
Completed | 189 | 204
Not Completed | 23 | 10
Period: Open Label Treatment Period (OLTP)
Arm/Group | DE-117 Ophthalmic Solution | Timolol Maleate Ophthalmic Solution 0.5%
Started | 377 (Some participants exited the study after Double Masked Treatment Period at Month 3, hence, 377 participants entered the Open Label Treatment Period.) | 0 (After completion of the Double Masked Treatment Period (DMTP), the adult participants converted to the single DE-117 QD arm at Month 3 to Open Label Treatment Period (OLPT) for additional 9 months.)
Completed | 304 (304 completed the study) | 0
Not Completed | 73 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Participants are similar in count to the Full Analysis Set Participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | DE-117 Ophthalmic Solution | Timolol Maleate Ophthalmic Solution 0.5% | Total
Number analyzed (Participants) | 212 | 213 | 425
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 7 | 13
  Between 18 and 65 years | 83 | 91 | 174
  >=65 years | 123 | 115 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (14.91) | 63.5 (14.48) | 64.1 (14.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 135 | 258
  Male | 89 | 78 | 167
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Black or African American | 48 | 52 | 100
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  White | 160 | 155 | 315
  Multiple | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 212 | 213 | 425

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure at Week 1
Description: Intraocular Pressure (IOP), the fluid pressure inside the eye was measured with calibrated Goldmann applanation tonometer in millimeters mercury (mmHg) at 3 time points throughout the day. Analysis using Mixed-Effects Model for Repeated Measures (MMRM)
Time Frame: 08:00, 10:00 and 16:00 at Week 1
Population: Full Analysis Set (FAS) included all randomized subjects who received at least one dose of study medication and provided baseline and at least one post-baseline IOP measurement. The number of analyzed are participants evaluable for the outcome measure at Week 1.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution | Timolol Maleate Ophthalmic Solution 0.5%
Number analyzed (Participants) | 212 | 213
mmHg
  8:00: number analyzed (Participants) | 210 | 211
  8:00 | 19.0 (0.22) | 19.1 (0.21)
  10:00: number analyzed (Participants) | 209 | 211
  10:00 | 18.0 (0.21) | 18.2 (0.21)
  16:00: number analyzed (Participants) | 211 | 210
  16:00 | 17.5 (0.21) | 17.9 (0.21)

2. Primary Outcome: Intraocular Pressure at Week 6
Description: as for outcome 1
Time Frame: 08:00, 10:00 and 16:00 at Week 6
Population: Full Analysis Set (FAS) included all randomized subjects who received at least one dose of study medication and provided baseline and at least one post-baseline IOP measurement. The number of analyzed are participants evaluable for the outcome measure at Week 6.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution | Timolol Maleate Ophthalmic Solution 0.5%
Number analyzed (Participants) | 212 | 213
mmHg
  8:00: number analyzed (Participants) | 202 | 208
  8:00 | 19.8 (0.20) | 18.4 (0.20)
  10:00: number analyzed (Participants) | 203 | 208
  10:00 | 18.9 (0.20) | 18.0 (0.20)
  16:00: number analyzed (Participants) | 201 | 208
  16:00 | 18.5 (0.21) | 17.7 (0.21)

3. Primary Outcome: Intraocular Pressure at Month 3
Description: as for outcome 1
Time Frame: 08:00, 10:00 and 16:00 at Month 3
Population: Full Analysis Set (FAS) included all randomized subjects who received at least one dose of study medication and provided baseline and at least one post-baseline IOP measurement. The number of analyzed are participants evaluable for the outcome measure at Month 3.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution | Timolol Maleate Ophthalmic Solution 0.5%
Number analyzed (Participants) | 212 | 213
mmHg
  8:00: number analyzed (Participants) | 196 | 203
  8:00 | 19.7 (0.24) | 18.5 (0.24)
  10:00: number analyzed (Participants) | 197 | 203
  10:00 | 18.8 (0.21) | 17.7 (0.21)
  16:00: number analyzed (Participants) | 196 | 203
  16:00 | 18.6 (0.22) | 17.8 (0.21)

4. Secondary Outcome: Mean Diurnal Intraocular Pressure (IOP) at Month 3 (First Key Secondary Endpoint)
Description: Mean Diurnal Intraocular Pressure (IOP) at Month 3: Analysis using Mixed-Effects Model for Repeated Measures (MMRM) on observed cases.
Time Frame: Month 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution | Timolol Maleate Ophthalmic Solution 0.5%
Number analyzed (Participants) | 196 | 203
mmHg | 19.0 (0.20) | 18.0 (0.19)

5. Secondary Outcome: Intraocular Pressure (IOP) at Week 1 With Baseline Mean Diurnal IOP Less Than 25 mmHg (Second Key Secondary Endpoint)
Description: Intraocular Pressure (IOP) at Week 1 with baseline mean diurnal IOP less than 25 mmHg (Second Key Secondary Endpoint)
Time Frame: 08:00, 10:00 and 16:00 at Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution | Timolol Maleate Ophthalmic Solution 0.5%
Number analyzed (Participants) | 140 | 138
mmHg
  8:00: number analyzed (Participants) | 139 | 136
  8:00 | 17.9 (0.25) | 18.2 (0.25)
  10:00: number analyzed (Participants) | 138 | 136
  10:00 | 17.2 (0.24) | 17.3 (0.24)
  16:00: number analyzed (Participants) | 139 | 135
  16:00 | 16.8 (0.25) | 17.2 (0.25)

6. Secondary Outcome: Intraocular Pressure (IOP) at Week 6 With Baseline Mean Diurnal IOP Less Than 25 mmHg (Second Key Secondary Endpoint)
Description: Intraocular Pressure (IOP) at Week 6 with baseline mean diurnal IOP less than 25 mmHg (Second Key Secondary Endpoint)
Time Frame: 08:00, 10:00 and 16:00 at Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution | Timolol Maleate Ophthalmic Solution 0.5%
Number analyzed (Participants) | 140 | 138
mmHg
  8:00: number analyzed (Participants) | 132 | 136
  8:00 | 18.7 (0.24) | 17.8 (0.24)
  10:00: number analyzed (Participants) | 133 | 136
  10:00 | 18.0 (0.25) | 17.4 (0.25)
  16:00: number analyzed (Participants) | 131 | 136
  16:00 | 17.6 (0.23) | 17.1 (0.23)

7. Secondary Outcome: Intraocular Pressure (IOP) at Month 3 With Baseline Mean Diurnal IOP Less Than 25 mmHg (Second Key Secondary Endpoint)
Description: Intraocular Pressure (IOP) at Month 3 with baseline mean diurnal IOP less than 25 mmHg (Second Key Secondary Endpoint)
Time Frame: 08:00, 10:00 and 16:00 at Month 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution | Timolol Maleate Ophthalmic Solution 0.5%
Number analyzed (Participants) | 140 | 138
mmHg
  8:00: number analyzed (Participants) | 129 | 133
  8:00 | 18.6 (0.29) | 17.7 (0.28)
  10:00: number analyzed (Participants) | 129 | 133
  10:00 | 17.8 (0.25) | 16.9 (0.25)
  16:00: number analyzed (Participants) | 129 | 133
  16:00 | 17.7 (0.25) | 17.2 (0.25)

8. Secondary Outcome: Mean Diurnal Intraocular Pressure (IOP) at Week 1 (Third Key Secondary Endpoint)
Description: Mean Diurnal Intraocular Pressure (IOP) at Week 1: Analysis using Mixed-Effects Model for Repeated Measures (MMRM) on observed cases.
  Mean Diurnal IOP at week 1 is defined as the average IOP of all three timepoints (8AM, 10AM and 4PM) at week 1.
Time Frame: Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution | Timolol Maleate Ophthalmic Solution 0.5%
Number analyzed (Participants) | 209 | 210
mmHg | 18.1 (0.19) | 18.4 (0.19)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent and were followed to resolution or until the subject's participation in the study ended for both Period 1 (Double Masked Treatment Period) at Month 3 and Period 2 (Open Label Treatment Period) at Month 12.
Description: Other Adverse Event data is a summary observed at a rate of 1.0% or higher by System Organ Class and Preferred Term for both the Double Masked and Open Label Periods.
  The summary of other adverse events in Double Masked Treatment Period and Open Label Treatment Period are independently summarized. For any other adverse events equal or over the threshold of 1% in open label but less than 1% in double masked, the AE will not be included in double masked (counted as 0). This is vice versa.
Groups:
- DE-117 Ophthalmic Solution (Double Masked Treatment Period): Topical DE-117 Ophthalmic Solution once daily and Vehicle once daily for 3 months for all subjects, followed by DE-117 Ophthalmic Solution once daily for additional 9 month for adult subjects only
  DE-117 Ophthalmic Solution: Topical DE-117 Ophthalmic Solution once daily and Vehicle once daily for 3 months for all subjects, followed by DE-117 Ophthalmic Solution once daily for additional 9 month for adult subjects only
- Timolol Maleate Ophthalmic Solution 0.5% (Double Masked Treatment Period): Topical Timolol Maleate Ophthalmic Solution 0.5% twice daily for 3 months for all subjects, followed by DE-117 Ophthalmic Solution once daily for additional 9 month for adult subjects only
  Timolol Maleate Ophthalmic Solution 0.5%: Topical Timolol Maleate Ophthalmic Solution 0.5% twice daily for 3 months for all subjects, followed by DE-117 Ophthalmic Solution once daily for additional 9 month for adult subjects only
- DE-117 Ophthalmic Solution (Open Label Treatment Period): Topical DE-117 Ophthalmic Solution once daily for 9 months for adult subjects only (Period 2)
Arm/Group | DE-117 Ophthalmic Solution (Double Masked Treatment Period) | Timolol Maleate Ophthalmic Solution 0.5% (Double Masked Treatment Period) | DE-117 Ophthalmic Solution (Open Label Treatment Period)
All-Cause Mortality (participants affected / at risk) | 0/211 | 1/215 | 1/377
Serious Adverse Events (participants affected / at risk) | 4/211 | 5/215 | 12/377
Other Adverse Events (participants affected / at risk) | 61/211 | 47/215 | 85/377
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DE-117 Ophthalmic Solution (Double Masked Treatment Period) (N=211) | Timolol Maleate Ophthalmic Solution 0.5% (Double Masked Treatment Period) (N=215) | DE-117 Ophthalmic Solution (Open Label Treatment Period) (N=377)
Cystoid macular (Eye disorders) | 1 | 0 | 3
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2
Influenza Type A test positive (Investigations) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Cerebral hemorrhage (Nervous system disorders) | 0 | 0 | 1
Acute Cardiac event (Cardiac disorders) | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DE-117 Ophthalmic Solution (Double Masked Treatment Period) (N=211) | Timolol Maleate Ophthalmic Solution 0.5% (Double Masked Treatment Period) (N=215) | DE-117 Ophthalmic Solution (Open Label Treatment Period) (N=377)
Conjunctival hyperaemia (Eye disorders) | 13 | 10 | 12
Vision blurred (Eye disorders) | 11 | 3 | 14
Photophobia (Eye disorders) | 10 | 1 | 4
Ocular hyperaemia (Eye disorders) | 6 | 4 | 0
Dry eye (Eye disorders) | 4 | 2 | 0
Eye pain (Eye disorders) | 4 | 5 | 6
Visual impairment (Eye disorders) | 4 | 0 | 0
Eye irritation (Eye disorders) | 3 | 8 | 4
Vitreous detachment (Eye disorders) | 3 | 1 | 0
Vitreous floaters (Eye disorders) | 3 | 0 | 6
Growth of eyelashes (Eye disorders) | 2 | 3 | 5
Macular oedema (Eye disorders) | 0 | 0 | 9
Cystoid macular oedema (Eye disorders) | 0 | 0 | 9
Punctate keratitis (Eye disorders) | 0 | 0 | 7
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 4
Eyelash changes (Eye disorders) | 0 | 0 | 4
Eyelash hyperpigmentation (Eye disorders) | 0 | 0 | 4
Eyelash thickening (Eye disorders) | 0 | 0 | 4
Sinusitis (Infections and infestations) | 0 | 0 | 5
Urinary tract infection (Infections and infestations) | 0 | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 4
Nasopharyngitis (Infections and infestations) | 0 | 4 | 0
Instillation site pain (General disorders) | 5 | 12 | 0
Vital dye staining cornea present (Investigations) | 7 | 5 | 8
Headache (Nervous system disorders) | 4 | 2 | 0
Hypertension (Vascular disorders) | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT03691649/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT03691649/SAP_001.pdf